CLINICAL TRIAL: NCT00523770
Title: An Exploratory Study in Healthy Elderly Subjects to Collect Urine for the Development of Assays to Detect Streptococcus Pneumoniae.
Brief Title: Exploratory Study in Healthy Elderly Subjects to Collect Urine for Development of Assays to Detect S. Pneumoniae
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: BACDU-001
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Infections, Streptococcal
Keywords: Invasive Pneumococcal Diseases; Pneumonia
MeSH Terms: conditions — Streptococcal Infections; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group A: Non-pneumococcal infected healthy elderly volunteers
  Interventions: Procedure: Urine sample collection

INTERVENTIONS:
Procedure: Urine sample collection — Urine samples will be collected and tested for the presence of S. pneumoniae

SUMMARY:
GSK Biologicals is working on the development of a vaccine to protect elderly people from pneumococcal infection. For the future studies in that project, it would be useful to have some easy non invasive tests to detect infection by the bacteria. Some tests on urine are already on the market but need to be improved in the laboratory. For that purpose, some urine samples from healthy subjects aged 65 years or above and who have not suffered from pneumonia nor have been administered pneumococcal vaccination in the past 3 months are needed.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 65 and 85 years of age at the time of the study.
* Written informed consent obtained from the subject
* Healthy subjects as established by medical history and clinical examination before entering into the study

Exclusion Criteria:

* Previous vaccination against Streptococcus pneumoniae in the 3 months before study start,
* History of pneumonia confirmed by documented radiology or any other diagnostic method within 3 months prior to study start

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Residents of Belgium and Finland
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-09; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Positive or negative result using Binax NOW S. pneumoniae Test | within one day

SECONDARY OUTCOMES:
Positive or negative result using the test to be developed for typing of S. pneumoniae | within one day
Positive or negative result using the test to be developed for detection of non-typable Haemophilus influenzae (NTHi) | within one day

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline